CLINICAL TRIAL: NCT02241239
Title: A Comparison of the Estimates of Fuwai and Reynolds Risk Model
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wuhan Asia Heart Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-0901-1
Record Dates: First submitted 2014-08-31; First posted 2014-09-16 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-08

CONDITIONS: Coronary Heart Disease and Stroke
MeSH Terms: conditions — Coronary Disease; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- participants: healthy adults without stroke and coronary heart disease

SUMMARY:
There are many risk prediction models. And their estimates are different. This study aimed to investigate the differences between the estimates of Fuwai and Reynolds risk model in Chinese, and investigate the reason for the differences.

DETAILED DESCRIPTION:
The participants will examined for cardiovascular risk factors, and their cardiovascular risks will be calculated based on the values of the risk factors using cardiovascular risk models. The estimates of different risk models will be compared, and the levels of traditional risk factors will be adjusted in order to evaluate the impacts of uncommon risk factors such as social and genetic risk factors.

ELIGIBILITY:
Inclusion Criteria: adults -

Exclusion Criteria: with coronary heart disease

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adults without coronary heart disease
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-08; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
cardiovascular risk | 1 day
  The cardiovascular risk is the probability of the occurrence of coronary heart disease and stroke. The cardiovascular risk is calculated by risk prediction models based on the patient's risk factors.

CONTACTS AND LOCATIONS:
Overall Officials: Youping Chen, M.D., Principal Investigator — Wuhan Asia Heart Hospital
Locations (2):
- China (2):
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - Wuhan Asia Heart Hospital, Wuhan